CLINICAL TRIAL: NCT01275716
Title: Impact of Coronary Images Used During Patient Education on Coronary Artery Disease and Subsequent Lifestyle Modifications. Is a Picture Really Worth a Thousand Words?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10-623-A
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease
Keywords: Patient Education; coronary artery disease; Impact of Coronary Images Used During Patient Education on Coronary Artery Disease and Subsequent Lifestyle Modifications.
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients who are shown the images (Experimental)
  Interventions: Behavioral: Impact of Coronary Images Used During Patient Education on Coronary Artery Disease and Subsequent Lifestyle Modifications
- Patients who are not shown the images (No Intervention)

INTERVENTIONS:
Behavioral: Impact of Coronary Images Used During Patient Education on Coronary Artery Disease and Subsequent Lifestyle Modifications — Subjects will be randomly assigned (like the flip of a coin) to a study group. One group will be given before and after treatment pictures of their affected heart arteries. The other group will not be shown these pictures. Both groups will still receive written and verbal information about living a heart healthy lifestyle and taking heart medications properly as part of their normal routine care.
  Arms: Patients who are shown the images

SUMMARY:
Subjects in this research study have Coronary Artery Disease (CAD). This occurs when there is a build-up of fatty material in the wall of the heart arteries that causes narrowing of the arteries. This could lead to chest pain, a heart attack, weakening of the heart and/or permanent damage to the heart. As part of their normal routine care, subjects had or will have a Percutaneous Coronary Intervention (PCI) to restore the blood flow in the arteries of their heart. During a PCI procedure, pictures are taken of the arteries before and after the treatment of the narrowing in the arteries. These pictures are acquired through angiography which is a way to produce X-ray pictures of the inside of arteries.

After a PCI procedure, there is a possibility for narrowing of the arteries to return. The likelihood of this happening can be greatly reduced by lifestyle changes and adhering to heart medication regimens. It is part of normal, routine care for CAD patients to be given written and verbal information on how to lead a heart healthy lifestyle and to take heart medications properly.

In this research study, the investigators will show half of the patients their before and after images of their heart arteries where the narrowing occurred and was treated. The other half of the patients will not be shown these images. Both groups will still receive information about lifestyle and medications as part of their normal, routine care. At the end of this study, the investigators will compare both groups to see if there are any differences in making lifestyle changes and taking heart medications properly. Additionally, the investigators would also like to see if there are any resulting differences in the amount of hearts attacks or other heart related medical events.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18
2. Able to provide informed consent in English.
3. Undergoing percutaneous coronary intervention for any clinical indication.

Exclusion Criteria:

1. Patients not able to provide informed consent.
2. Patients without a means for telephone communication.
3. Incarcerated individuals and other special populations.
4. Patients unable to or unwilling to reliably participate in telephone followup.
5. Significant neurologic co morbidities such as cerebrovascular accidents with deficit or developmental delays which may impact learning and/or memory
6. Any medical comorbidity which might result in life-expectancy < 1 year
7. Any other condition of sufficient severity to impair cooperation in the study- i.e. substance abuse, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-26 (Actual)

PRIMARY OUTCOMES:
Significant improvement of patient's knowledge in the group that receives the images versus the group that receives standard education of coronary artery risk factors as measured on questionnaires from baseline to 30 days and at 3 and 6 month follow up | 6 months

SECONDARY OUTCOMES:
The secondary endpoints of the study is a significant improvement in the patient's adherence to nutritional, exercise and medical regimen in the group receiving the images and education versus the group that receives standard education alone | 6 months
An exploratory analysis will assess the impact of the aforementioned educational intervention on the occurrence of major adverse cardiovascular events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Nathan, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States